CLINICAL TRIAL: NCT07231146
Title: Interaction Between Milk and Yogurt and Gastrointestinal Hormone Response on Cognitive Performance in School-Aged Children
Brief Title: Interaction Between Dairy and Gut Hormone Response on Cognitive Performance in Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: National Dairy Council (Other); Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Nick Bellissimo, PhD, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB 25-066
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Children; Healthy
Keywords: Cognitive Performance; Dairy; Gastrointestinal Hormones; Emotions; Mood
MeSH Terms: interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Fat-Free Milk Treatment (Experimental): Test Treatment
  Interventions: Other: Fat-Free Milk
- Low-Fat Milk Treatment (Experimental): Test Treatment
  Interventions: Other: Low-Fat Milk
- Full-Fat Milk Treatment (Experimental): Test Treatment
  Interventions: Other: Full-fat Milk
- Snack Skipping Treatment (Experimental): Test Treatment
  Interventions: Other: Snack Skipping
- Fat-Free Yogurt (Experimental): Test Treatment
  Interventions: Other: Fat-Free Yogurt
- Low-Fat Yogurt (Experimental): Test Treatment
  Interventions: Other: Low-Fat Yogurt
- Full-Fat Yogurt (Experimental): Test Treatment
  Interventions: Other: Full-Fat Yogurt

INTERVENTIONS:
Other: Fat-Free Milk — Fat-free milk (500 mL, skim, 0%, Lactantia PurFiltre) will provide 180 kcal, 0.4 g fat, 26 g carbohydrate, and 18 g protein. Treatments matched for calories (180 kcal).
  Arms: Fat-Free Milk Treatment
Other: Low-Fat Milk — Low-free milk (346 mL, 2%, Lactantia PurFiltre) will provide 180 kcal, 6.9 g fat, 16.6 g carbohydrate, and 12.5 g protein. Treatments matched for calories (180 kcal).
  Arms: Low-Fat Milk Treatment
Other: Full-fat Milk — Full-free milk (281 mL, 3.25%, Lactantia PurFiltre) will provide 180 kcal, 9.0 g fat, 13.5 g carbohydrate, and 10.1 g protein. Treatments matched for calories (180 kcal).
  Arms: Full-Fat Milk Treatment
Other: Snack Skipping — Snack skipping (no caloric contribution).
  Arms: Snack Skipping Treatment
Other: Fat-Free Yogurt — Fat-free Yogurt (242.3 g, Oikos High Protein Vanilla; 0% MF) will provide 180 kcal, 0 g fat, 20.8 g carbohydrate, and 23.5 g protein. Treatments matched for calories (180 kcal).
  Arms: Fat-Free Yogurt
Other: Low-Fat Yogurt — Low-fat Yogurt (210.0 g, Oikos Original 2% MF) will provide 180 kcal, 3.6 g fat, 21.6 g carbohydrate, and 15.6 g protein. Treatments matched for calories (180 kcal).
  Arms: Low-Fat Yogurt
Other: Full-Fat Yogurt — Full-fat Yogurt (185.3 g, Oikos Extra Creamy Vanilla 9% MF) will provide 180 kcal, 15.9 g fat, 21.2 g carbohydrate, and 6.4 g protein. Treatments matched for calories (180 kcal).
  Arms: Full-Fat Yogurt

SUMMARY:
The purpose of this study is to investigate the short-term effects of milk and yogurt of varying fat and protein content on cognitive performance in healthy children aged 9 - 14 years; and to provide insight into mechanisms by which dairy consumption may affect cognitive performance through gastrointestinal (GI) hormone responses. The investigators hypothesize that the consumption of dairy products, specifically their protein and fat components, will improve cognitive performance via its interaction with the gut-brain axis in children. Furthermore, the investigators hypothesize that all milk and yogurt products will enhance cognitive performance over 120- mins compared to snack skipping through its interaction with GI hormones, with a greater effect in higher fat containing milk and yogurt products.

DETAILED DESCRIPTION:
A randomized within-subject repeated measures experiment will be used to study the effect of milk and yogurt of varying fat content on cognitive performance and its interaction with GI hormones in children (9-14 years). Participants will consume milk [Experiment A] and yogurt [Experiment B] test treatments, followed by measures of cognitive performance, blood glucose and GI hormone biomarkers over 120-min. In Experiment A and B, participants will consume, in a random order on separate mornings, one of four test treatments: (1) Full-fat, (2) Low-Fat, (3) No-fat, and (4) Snack-skipping test treatments. Cognitive domains (learning and memory, spatial working memory, attention, processing speed, and executive function), gastrointestinal hormone response, and subjective emotions will be assessed at baseline (0-min), and 30-, 60-, and 120-min following treatment consumption.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 14 years of age;
* Normal weight is defined as being between the 5th and 85th percentile for age and biological sex at birth according to the Centers for Disease Control growth reference charts

Exclusion Criteria:

* Children with overweight/ obesity;
* Children with food sensitivities or allergies to dairy, gluten or any foods used in the study;
* Children with any diagnosed learning, emotional, or behavioural disabilities;
* Children taking any medications that may influence cognitive performance.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Learning and short-term memory | Immediate measured at 30-minutes post-treatment and delayed at 60- and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Learning and short-term memory will be assessed using an immediate and delayed Word Recall Test (accuracy).
Spatial working memory | Change from baseline (measured at 0-minutes before treatment) and at 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Spatial working memory will be assessed using the forward and backward versions of the Corsi Block Test (accuracy).
Sustained Attention | Change from baseline (measured at 0-minutes before treatment) and at 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Sustained attention and processing speed will be assessed using the Continuous Performance Test (CPT) (accuracy).
Executive Function | Change from baseline (measured at 0-minutes before treatment) and at 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Executive function and selective attention will be assessed using the Flanker Task (accuracy)

SECONDARY OUTCOMES:
Subjective mood and emotion | Change from baseline (measured at 0-minutes before treatment) and at 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  A visual analogue scale (VAS) with twelve questions will be administered to assess subjective emotions and mood (aggression, anger, excitement, disappointment, happiness, upset, frustration, alertness, sadness, tension, calmness, sleepiness, and wellness). Individual questions will be used to form a composite emotion score. Each VAS will be administered via a digital software application (Express VAS, Toronto, Ontario, Canada) on a Dell tablet where children will place an 'X" on the VAS line (100 unit scale) to describe their feelings.
Gastrointestinal Hormone Response | Change from baseline (measured at 0-minutes before treatment) and at 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Blood biomarkers will include glucose, insulin, active GLP- 1, and total GIP. Blood samples will be collected via a venous catheter inserted into the participants arm by a Registered Nurse

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No